## UNIVERSITY OF PENNSYLVANIA RESEARCH SUBJECT INFORMED CONSENT AND HIPAA AUTHORIZATION FORM

| Protocol Title: | Open-labeled trial of Zepatier for treatment of hepatitis C negative patients who receive heart transplants from hepatitis C positive donors (USHER) |
|---|---|
| Sponsor: | University of Pennsylvania |
| Funder: | Merck & Co. |
| Principal Investigator: | David Goldberg, MD, MSCE<br>(215) 746-8598 |
| Co-Principal<br>Investigator: | Peter Reese, MD, MSCE<br>(215) 900-3782<br>Rhondalyn Forde-McLean, MD, MHS<br>(215) 662-2727 |
| Study<br>Coordinator: | Anna Sicilia, BS<br>(215) 746-7105 |
| Emergency<br>Contact: | 24 Hour Emergency Numbers Dr. Reese: (215) 900-3782 Dr. Goldberg: (646) 242-6349 (215) 662-6200 - Ask for Heart Transplant Coordinator on Call |

## Why am I being asked to volunteer?

You are being asked to participate in this trial because you are expected to have 6-12 months, or more, before you receive a heart transplant.

We are asking you to consider joining a study where hearts with hepatitis C will be offered to people like you who do not have hepatitis C. Hepatitis C is a virus that infects your liver, and over many years (10-30), can lead to scarring of your liver, which can develop into end-stage scarring (called cirrhosis), which could lead to liver failure, cancer, or death. Rarely, hepatitis C can cause inflammation in other parts of your body, including your skin or kidneys.

If you receive a heart with hepatitis C, we would give you free medicine to treat the hepatitis C virus. The treatments for hepatitis C are highly effective. In other studies, these medicines have cured more than 95% of patients with chronic hepatitis C. However, we do not know whether these medicines will be as effective for someone who becomes infected with hepatitis C after a heart transplant.

Your participation is voluntary which means you can choose whether or not you want to participate. If you choose not to participate, your care at Penn and your priority on the

heart transplant waiting list will not change. You will receive the usual care for someone on the transplant waiting list.

Before you can make your decision, you will need to know what the study is about, the possible risks and benefits of being in this study, and what you will have to do in this study. The research team is going to talk to you about the research study, and they will ask you to read this consent form carefully. You may also decide to discuss it with your family, friends, or family doctor. You may find some of the medical language difficult to understand. Please ask the study doctor and/or the research team about this form. If you decide to participate, you will be asked to sign this form.

## What is the purpose of this research study?

Currently there are over 4,000 people waiting for a heart transplant in the United States, but there are only about 2,800 heart transplants from deceased donors performed each year. Because there are not enough hearts available for all the people who need them, average waiting times for heart transplantation can be more than 6-12 months, especially for patients with blood types A, B, or O, or for patients who are "bigger" (either height or weight).

One potential option to increase the number of available hearts is to allow patients without hepatitis C to accept a heart from a donor with hepatitis C. In almost all cases, hearts from donors with hepatitis C are not given to patients without hepatitis C.

The purpose of this study is to determine whether it is safe to give recipients without hepatitis C, a heart from a donor with hepatitis C. Additionally, this study will evaluate whether treatments given after transplant, can cure hepatitis C in individuals who receive hearts from donors with hepatitis C.

In this study, recipients who receive a heart infected with hepatitis C will be treated with a pill made of Grazoprevir + Elbasvir (Zepatier) after the transplant. These two medications are combined in one pill that has recently been approved by the FDA in the US for the treatment of chronic hepatitis C in adults.

This study is funded by Merck, the company that makes Zepatier.

# How long will I be in the study? How many other people will be in the study?

Participants will be in the study while they wait for a heart transplant (estimated to be ~3-6 months but could be shorter or longer) and for approximately 1 year after they get a heart transplant to allow us to follow-up the subjects' health before and after transplant. Upon receiving a heart transplant from a hepatitis C-positive donor, subjects will be followed until their hepatitis C level is positive. Treatment will commence, with the hepatitis C treatment duration between 12 and 16 weeks depending on the exact HCV subtype.

This study will enroll around 30 patients at the Hospital of the University of Pennsylvania (HUP). Of those 30, we anticipate that ten patients will receive a heart transplant with hepatitis C. We believe that all the patients who get a transplant will become infected with hepatitis C virus and therefore need treatment for hepatitis C virus.

## What am I being asked to do?

Your participation in the study involves multiple visits to the Hospital of the University of Pennsylvania over a period of up to 6 months after heart transplant (each study visit will usually coincide with a regular post-heart transplant visit), and an additional visit 12 months after your heart transplant. While you are on the waiting list, we will also monitor your health. Many of these visits will require collection of blood to be used for safety labs (such as blood counts and liver tests), as well as labs to determine the amount of hepatitis C virus in your blood (hepatitis C viral load), and special ultrasound tests to measure how stiff your liver is.

## This study involves three (3) phases:

### Phase 1: Screening

The screening period is the period of time when it is determined if you are eligible to be in the study. This will take place before you receive a heart transplant with hepatitis C and before you begin treatment with the study drug. During screening, you will review and sign this consent prior to any study procedures. Some of the exams, tests, or procedures may have already been done as part of your routine care. If you have had some of these tests done already, they may not need to be repeated. This decision will be up to your study doctor. The screening procedures may take up to 5 hours and includes the following:

- A complete physical exam
- Review medications
- Assessment of current health status
- Blood sample collection
  - to measure blood counts and to test the function of your organs such as your hearts and liver
  - for a pregnancy test (for women who are able to have children)
  - for research purposes (this may include tests to your immune responses)

## Phase 2: Waiting List

Following screening, if you are determined to be eligible for the study, we will change your transplant records to show that you are willing and eligible to receive offers for hearts from donors with hepatitis C. You will remain on the heart transplant waiting list. During that time, you will still be able to receive offers of hearts from donors without hepatitis C.

If you do get an offer of a heart with hepatitis C, we will test the donor to see what hepatitis C genotype the donor has. We are only accepting hearts from donors that have hepatitis C genotype 1 and 4, because this type of hepatitis C virus is easier to treat. The test for hepatitis C genotype is not perfectly accurate, although studies have shown that it is >95% accurate. However, all genotypes of hepatitis C can be treated, although some genotypes are more difficult to treat than others (although with current available therapies, cure rates of ≈90% can be achieved with all genotypes).

If you do get an offer of a heart, you can decide with your doctor whether or not you want to accept the heart.

If you do not get a heart transplant from a donor with hepatitis C during the study period, or if you get a heart transplant without hepatitis C, then you will not need any study related treatments or treatment-related study visits. We will review your medical records to monitor your health.

If you do get a heart transplant with hepatitis C, then you will need to come to study visits that take place the same day as your regular visit with your doctor. We will closely monitor your health. If we detect hepatitis C virus in your blood, then we will treat you for the infection. Then you will enter Phase 3 of the study, which we describe next.

## Phase 3: Transplantation

We will monitor your blood for hepatitis C infection. It is possible that some people who are infected with hepatitis C from a heart transplant will be able to rid themselves of the virus through their own immune system. However, we expect that almost everyone in the study who receives a hepatitis C infected heart transplant will become chronically infected with the virus. We will begin treatment for hepatitis C as soon as we detect the virus in your blood.

### Study Drug

After transplantation, study participants with hepatitis C will receive 12 weeks of Zepatier treatment. The study drug includes Grazoprevir + Elbasvir and is given as a single combination pill each day. We will supply enough study drugs at each visit to last until your next visit. Also, prior to starting the medication, we will check to see if there are mutations in the virus. If by chance certain mutations are found, your treatment may be lengthened to 16 weeks, instead of the original 12 weeks, in addition to receiving an additional medication, Ribavirin, if your heart function allows for it.

If by chance your hepatitis C is not cured after receiving Zepatier for 12 weeks, then you will be provided with a second treatment that includes Zepatier, plus 2 additional medications which have been used to treat Hepatitis C (Sofosbuvir and Ribavirin) to try to cure your hepatitis C infection.

Zepatier works by blocking the hepatitis C virus from multiplying in your body. In studies of patients with hepatitis C who had not received a heart transplant, cure rates using these medications have been over 95%.

The drug will be provided by the manufacturer who is sponsoring the study.

The cure rate of Zepatier has not been established in patients who undergo heart transplantation and become infected with hepatitis C from the heart. The safety and tolerability of Zepatier after heart transplantation have also not been studied. However, in the event dialysis is needed after your transplant due to acute kidney injury, we do know that the cure rates for patients with known hepatitis C and chronic kidney disease (including being on dialysis) are similar to rates of patients without kidney disease.

Zepatier has been approved by the Food and Drug Administration. This drug regimen was chosen as first-line therapy for this study rather than other approved agents because this investigational agent is unique in that it can be safely used in patients with abnormal heart function. As a result, if your heart function has not fully recovered when treatment is initiated after transplant, the investigational agents can be safely given to you.

### Other Medications

You will continue to take all the other medications prescribed by your doctor during the study. Your medication list will be reviewed during the screening visit and approved if you are eligible for the study. It is extremely important to provide an accurate list of all your medications (prescribed, over-the-counter, and herbal) at each visit and to take them as directed. However, we will not supply other medications.

**Study Visits 1 – 4:** The first visit will take place in the hospital during your recovery from surgery. Visits 2 – 4 will take place approximately every week - on the same days as your heart transplant clinic visits.

Someone from the research team will attempt to contact you before each appointment to remind you where to go and relay any special instructions.

During these visits, the following may be performed:

- Phlebotomy (drawing a blood sample), to measure for presence of the hepatitis C virus and to test the virus for mutations (NS5A Resistance Testing) that would lead to longer treatment.
  - NS5A Resistance testing is a type of blood test to check for mutations in the virus. This test is not approved by the Food and Drug Administration (FDA), but is validated by the Clinical Laboratory Improvement Amendments (CLIA). CLIA is a certification that allows clinical laboratory results to be shared with patients. This test is part of routine clinical care, and it is "recommended" by the FDA to be used to help guide treatment decisions in patients with genotype 1a (a subtype of genotype 1) hepatitis C who are being treated with Zepatier.
- Talk to you about how you feel and perform a physical examination, if necessary

Review your medications

If your blood tests show hepatitis C in your blood, we will call you and make arrangements for you to start treatment for hepatitis C. We will also notify your medical team that you are beginning treatment for hepatitis C.

**Study Visits 5 – 9:** These visits will take place every two to four weeks - on the same days as your heart transplant clinic visits.

Someone from the research team will attempt to contact you before each appointment to remind you where to go and relay any special instructions.

You may receive phone calls from research staff in between appointments to confirm that you are taking the study drug as prescribed.

The following procedures may be performed:

- Obtain blood samples to measure for presence of the hepatitis C virus
- Talk to you about how you feel and perform a physical examination, if necessary
- Review your medications
- Assess side effects and potential adverse events
- Count study pills and review drug diary for compliance
- Provide additional study pills

**Research blood samples:** Throughout the study, we will collect blood samples to measure for presence of the hepatitis C virus. This will be coordinated with blood tests for the transplant team.

**Additional visits:** These will only be necessary if the treatment does not cure you of hepatitis C. In that case, we will provide you Zepatier for an additional 12 weeks, and add two other hepatitis C medications (Sofosbuvir and Ribavirin), provided by the study investigators. These additional medications should increase the chance of curing you of hepatitis C.

### Follow-Up Period

The Follow-up Period is after you have stopped taking the study drug. It is important that you return for all follow-up visits so that your health can be reviewed.

**Study Visit 10:** This will be about 6 months after your transplant. The following procedures may be performed:

- Obtain blood samples
- Review your medications
- Assess side effects and adverse events
- Assess current health status
- Transient elastography (FibroScan®)

During this visit, your study results will be discussed with you, and as your test results become available, someone from the study team will keep you up to date on the status of your hepatitis C infection, after treatment

**Study Visit 11:** This will be about 12 months after your transplant. The following procedures may be performed:

- Obtain blood samples
- Review you medications
- Assess current health status
- Transient elastography (FibroScan®)

## What are the possible risks or discomforts?

The main risk of this study is that you will become infected with hepatitis C. The main potential benefit of this study is that you could get a heart transplant sooner than if you only accept offers of hearts from donors without hepatitis C infection.

## 1. Risks related to transplantation with a hepatitis C heart

### Liver problems

You should know that it is possible that the treatment for hepatitis C will not work as well after a transplant as it has worked in patients who do not have a transplant. It is also possible that after heart transplant, a hepatitis C infection could cause you serious health problems, including liver failure or death. Hepatitis C can rarely cause severe liver inflammation in the first few weeks to months after infection, or the virus can cause scarring and failure of your liver over many years.

In the short term, infection with hepatitis C can cause a flu-like illness that includes fatigue, nausea, fever, abdominal pain, vomiting, joint pain, and jaundice (yellow skin). In very rare circumstances, acute infection with hepatitis C can cause severe inflammation or even liver failure, including a condition called fibrosing cholestatic hepatitis. The risk of this complication in patients without hepatitis C who receive a transplant from a donor with hepatitis C is unknown. This complication can be treated and cured in some cases with the medications the investigators will be providing.

Liver failure can cause someone to experience leg swelling, yellow skin, uncomfortable feelings of itchiness, bleeding, breathing problems and the abdomen to fill with fluid. Liver failure can also cause death. Based on the limited data available, we believe that it would be rare for someone in the study to experience liver failure in the first months after transplantation, when we would give treatment. However, because liver failure is possible, we are only enrolling individuals in this study who would potentially be eligible to receive a liver transplant if they developed liver failure after a heart transplant, in addition to a clinical evaluation by a liver doctor (hepatologist) and liver transplant surgeon, which are not required for a heart transplant.

If your hepatitis C cannot be cured with the first-line and second-line treatments through this trial, over many years, there may be continued inflammation and scarring

of your liver that over many years can lead to cirrhosis and eventually liver failure. Longer term infection with hepatitis C increases the risk of developing liver cancer, liver failure requiring a liver transplant, or death.

## Additional risks of hepatitis C:

Hepatitis C can cause other types of inflammation in your body, such as arthritis, rash, anemia and inflammation damage to your heart transplant. However, these problems should respond to effective treatment for the virus.

There may also be a small risk of developing Focal and Segmental Glomerulosclerosis (FSGS) after receiving a kidney from a donor with hepatitis C. FSGS is a disease that harms the filters of the kidney and causes a patient to lose protein in their urine. However, this condition can also develop in patients who do not have hepatitis C. Long term, FSGS may cause kidney failure. After transplant, we will monitor all patients for conditions like FSGS. We will also offer treatments for FSGS, which can help some patients.

## Risks of the test used to determine the hepatitis C virus genotype

In this study, we intend only to transplant organs from patients with a certain type of hepatitis C – genotype 1. This type of the virus is easier to cure. There is less than a 1% chance that the test we use to identify the virus might not be 100% accurate. If the test gives the wrong result and you get a heart that has a different genotype of virus in it, your chances of being cured may be lower.

## 2. Risks related to study medication

### Side effects from medication:

When receiving treatment for hepatitis C, you may have side effects. Everyone taking part in the study will be watched carefully for any side effects. Side effects may be mild or serious. You should talk to your study doctor about any side effects that you experience while taking part in the study. If you are injured for any reason while you are in the study, you should tell the treating doctor or hospital that you are taking part in the study.

### Side Effects of Zepatier

There is a risk of serious and/or life-threatening side effects when non-study medications are taken with the study drug. For your safety, you must tell the study doctor or nurse about all medications you are taking before you start the study drug and also before starting any new medications while in the study. Also, you must tell the study doctor or nurse before enrolling in any other clinical trials while in this study.

In studies, this drug has been generally well tolerated. Risks and side effects related to Zepatier include:

## Most Common

1) Feeling tired or weak, 2) Headache

#### Less Common

3) Nausea, 4) Diarrhea, 5) Insomnia, 6) Joint soreness, 7) Itching, 8) Rash,

9) Shortness of breath, 10) Anemia (low red blood cell count)

#### Rare

11) Abnormal liver function tests suggesting liver inflammation, 12) Abnormal pancreas function tests suggesting pancreas inflammation, 13) depression, 14) abdominal pain, 15) irritability

Tell your healthcare provider right away if you get any of the following symptoms or if they get worse during treatment with Zepatier:

- loss of appetite
- yellowing of your skin or eyes
- nausea and vomiting
- color changes in your stool
- feeling tired or weak

There may be other side effects that have not yet been described including severe allergic reaction. It is also possible that taking medications to prevent your immune system from rejecting your heart transplant (also known as immunosuppression) at the same time as Zepatier might change its effectiveness or side effects.

## **Resistance of the virus to hepatitis C treatments:**

We do not know how effective Zepatier will be in eliminating hepatitis C after a transplant, in your circumstances. Determining the medication's effectiveness is one of the purposes of our study. One of the main risks of participating in this study is the possibility that hepatitis C may become resistant to the medication and may limit your future treatment options. The likelihood of resistance developing is higher if you skip doses or do not follow the study recommendations. If you show possible resistance to the study drug by having an increase in your hepatitis C viral load while on treatment, you will be asked to return to repeat the hepatitis C viral load test quickly. We may change your treatment plan.

Very few people (approximately 5%) have a mutation of a type of hepatitis C that puts them at risk for resistance. We will conduct a test to determine if you are at risk for this. As with the genotyping test, there is a risk that the test is not 100% accurate. If the test gives the wrong result, your chances of being cured may be lower and you may need additional treatment.

If you do not respond to treatment with Zepatier after 12 weeks, we will offer you a different set of medications (Sofosbuvir and Ribavirin) in addition to another round of Zepatier to treat your hepatitis C. It is unknown if this alternative set of medications will succeed in curing you of hepatitis C, although the expectation of the investigators is that it will likely be successful in curing you of your hepatitis C.

Risks and side effects related to the additional use of Sofosbuvir and Ribavirin include:

Most Common

1) Feeling tired or weak, 2) Headache, 3) Nausea/stomach pain, 4) Anemia, 5)

Insomnia,

6) Rash, 7) Itchiness, 8) Shortness of breath

### Less Common

9) Cough, 10) Dry skin, 11) Diarrhea, 12) Vomiting, 13) Low appetite, 14) Indigestion, 15) Sore muscles, 16) Feeling irritable/depressed, 17) Sore joints, 18) Nasal irritation, 19) Abnormal liver function tests, 20) Abnormal pancreas function tests, 21) Low white blood cell counts, which can increase vulnerability to infection, 22) Low platelet counts, which can increase vulnerability to bleeding, 23) birth defects from Ribavirin when either the man or woman is currently taking Ribavirin at the time of contraception, or had used Ribavirin in the preceding 6

## 3. Risks related to study procedures and tests Blood Drawing

The potential risks of the needle stick to draw blood include pain, bruising, bleeding, fainting, and infection. Discomfort from this procedure is generally short lasting, and serious side effects are extremely rare. Some people experience feelings of lightheadedness or dizziness after having blood drawn. The amount of blood drawn will be within the limits allowed for adult participants.

### **Genetic Testing**

months.

Some of the blood drawn from you as part of this study will be used for genetic tests. Genetic tests can help researchers learn about potential relationships between response to HCV treatment and genetic factors. Human leukocyte antigen (HLA) testing will also be completed. This is a genetic test of markers of the immune system.

We will not release any information about you or your family to relatives, any insurance company, employer, or your primary care physician without your written permission. There may be a risk that genetic information obtained as a result of participation in research could be misused for discriminatory purposes. However, state and federal laws provide some protections against genetic discrimination. Researchers who will have access to genetic information about you will take measures to maintain the confidentiality of your genetic information. Although we are committed to confidentiality, a court could still subpoena your medical records. All of these issues should be carefully considered before joining the study.

#### Risk of Stored Samples (Optional)

If you agree to have samples stored for future research use, there may be confidentiality risks associated with the storage and analysis of your samples or the information resulting from the analysis of your samples. For example, if future research involves genetic testing there's a potential risk associated with the release of private health information, though every effort will be made to maintain your confidentiality.

## Discovery of health problems during screening

During screening for this study, we will examine you and perform studies as apart of screening. It is possible that by doing these studies, we will identify new health

problems that you weren't aware of. If we discover new health problems, we will answer your questions and try to arrange appropriate treatment if any is needed. If new health problems are discovered, it is possible that you would not be able to enter this study. It is also possible that you would no longer be eligible for heart transplantation based on the results.

## Reproductive risks

If you do become pregnant, Zepatier may cause problems to your fetus. The risks to a fetus or a nursing child are not known at this time, so women who are pregnant or nursing a child may NOT join the study.

All <u>women</u> who can have children must have a test that shows they are not pregnant before the study drug is given and will be counseled regarding the importance of avoiding pregnancy during study treatment, including the use of highly effective methods of birth control. Women who can have children must engage in a highly effective form of birth control while in the study and six weeks afterwards. We define highly effective birth control the same way that the transplant program does. Notably, the use of transplant anti-rejection drugs can cause birth defects.

### Examples include:

- 1) sexual abstinence, or
- 2) a vasectomized partner, or
- 3) an intrauterine device (IUD), or
- 4) a hormonal method such as oral contraceptive pill PLUS a barrier method such as a condom, or
- 5) Diaphragm with spermicide PLUS a condom

Even if you use birth control there is a small chance that you could become pregnant. If you suspect that you have become pregnant, you must notify the study doctor immediately. If you become pregnant during the study, it is important that you tell us right away.

<u>All men and women</u> in the study who are sexually active must ALSO use a barrier method of contraception – such as condoms - while they are in the study and while they have hepatitis C. Although it is rare, hepatitis C can sometime be spread through sex. Barrier contraception during *any* sexual activity is important to keep your partner from getting infected with the virus.

<u>All men and women</u> who require Ribavirin therapy will be required to use two forms of contraceptive therapy while on Ribavirin therapy, and for up to 6 months after the last dose of the study drug due to the risk of birth defects from the use of Ribavirin. Men are required to also use birth control because Ribavirin can affect the sperm in a manner that can lead to birth defects.

## What if new information becomes available about the study?

In addition to the risks described above, there may be unknown risks, or risks that were not anticipated, associated with being in this study. If new information becomes available about the study drug that might affect your willingness to continue participation your study doctor will inform you immediately and will discuss with you whether you want to continue to participate in the clinical study.

You may be asked to sign a revised consent form if this occurs. You have the right to decide either to continue with the clinical study or to withdraw.

## What are the possible benefits of the study?

The main benefit of the study is that you may receive a heart transplant earlier than you would have if you chose to wait for a heart without hepatitis C. Receiving a heart transplant earlier will lead to clinical benefits as your heart function improves as well as improve your quality of life. Also, receiving a heart may increase your overall lifespan by decreasing your risk of dying while waiting for a transplant.

## What other choices do I have if I do not participate?

We encourage you to discuss this study with your physician and to explore other treatment options. Other treatment options include not enrolling in this study and waiting for a heart transplant from a heart donor who does not have hepatitis C.

However, if you decide not to join the study, you may instead remain on the waitlist for a longer period of time and suffer health consequences, including death or additional complications.

## Will I be paid for being in this study?

You will not receive any form of payment for your participation in this study.

## Will I have to pay for anything?

The heart transplant itself will be paid for by your insurance carrier, and does not require any additional pre-authorization because of the potential to receive a heart from a hepatitis C-positive donor. The costs of all visits and tests described above will be billed to you or your insurance carrier, except for the blood draw for research purposes (which includes the hepatitis C genotype test which is based on a laboratory-developed test using materials purchased from the commercial entity that developed this test, and will be paid for by the research team), and the study drug, which will be paid for by the study funder. You are still responsible for any deductibles or applicable co-pays for routine office visits, blood work and procedures. Please talk to your doctor and study team about putting you in touch with a financial counselor to determine exactly what the deductible and co-pay will be for you; this is highly variable depending on your type of insurance.

## What happens if I am injured from being in the study?

If you become sick or injured as a direct result of taking the study product(s) the Hospital of the University of Pennsylvania will provide you with medical treatment. The Sponsor, the University of Pennsylvania, will reimburse you for the reasonable and necessary costs of such medical treatment. No other form of reimbursement for study-related injury or illness is offered by the Sponsor. You should immediately contact your Study Doctor at the contact information shown on the first page of this form, in the event you experience any study-related illness or injury.

If you receive Medicare benefits, the Sponsor, the University of Pennsylvania, is required by law to report payments made to you for treatment, complications, and injuries that arise from this Study. Information that you are taking part in the Study, medical treatments received, Medicare claims, and other personal information about you such as your name, social security number, and date of birth, will be provided to the Centers of Medicare and Medicaid Services and its agents and/or contractors for this purpose.

You do not give up your legal rights by signing this form.

If you think you have been injured as a result of taking part in this research study, tell the person in charge of the research study as soon as possible. The researcher's name and phone number are listed at the beginning of the consent form.

We are committed to offering you with treatment for hepatitis C infection during the study. We expect that these treatments are likely to cure you of the infection. However, it is possible that treatment will not cure the infection and that you would develop health complications. Once the study ends, we would expect you to seek appropriate treatments for hepatitis C infection through your insurance or private means.

## When is the Study over? Can I leave the Study before it ends?

This study is expected to end after all participants have completed all visits, and all information has been collected. Tell the study doctor if you are thinking about stopping or decide to stop. He or she will tell you how to stop your participation safely. It is important to tell the study doctor if you are thinking about stopping so that your doctor can evaluate any risks and discuss what alternative follow-up care and testing could be most helpful for you.

### Reasons for Stopping Study Medication

If you are not responding to the study medication (checked frequently by measuring the levels of hepatitis C in your blood) or develop a potential life threatening complication from the medication, we will stop the study medications completely. However, you will still be followed but less frequently. Regardless of the stage of liver disease, the recommendations are to treat hepatitis C if medically possible, however some physicians might choose to wait and not treat in the immediate future.

### Reasons for Withdrawal or Study Discontinuation

Your involvement in this study is entirely up to you. You may leave the study at any time and for any reason. Withdrawal will not interfere with your future care. If you decide to leave, we may ask you to return for a final visit to perform tests and exams to ensure safety. However, you will not be required to return for this visit.

You may be discontinued from the study (taken off the study without our asking for your permission) if:

- You become pregnant while undergoing treatment with Zepatier. Therapy will be stopped as there are no safety data of Zepatier during pregnancy. Patients will continue with the regularly scheduled study visits, but will not be eligible to receive continued Zepatier therapy.
- We cannot locate you, or if you miss multiple visits or study drug doses.
- You develop a condition that it is life threatening or any other significant risk as judged by the Investigators.
- We or your primary care provider believe that it is in your best interest to stop taking the study medications even if the criteria required for stopping treatment have not been met.
- Zepatier is no longer produced by the company, or if a decision is made to stop the study.

# Who can see or use my information? How will my personal information be protected?

Your medical records will be kept confidential to the extent allowed by the law. Your name or any other data that might identify you will not be used in any reports or publications resulting from this study. Because of your consent to participate, your medical records may be reviewed by the study Sponsor and by Penn's Institutional Review Board (the group that is responsible for making sure that the study follows the guidelines for the protection of human research subjects) with the understanding that these records will be used only in connection with carrying out obligations relating to this clinical study. We will also give information about you to your personal doctors. You may change doctors whenever you like, but we need to have a doctor with whom we can communicate about you. We would not ask your permission for each of these contacts.

Data from this study will be entered into a computerized database through a secured website. Only authorized personnel using a password will be permitted to enter and access data. You will not be identified by name, social security number, or medical record number in the study database. Each patient will be assigned a unique study ID code for identification. Records linking the study ID code with any personal identification information will be kept by the study team in a locked area.

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a> as required by the U.S. Law. This web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this web site at any time.

## Electronic Medical Records and Research Results What is an Electronic Medical Record?

An Electronic Medical Record (EMR) is an electronic version of the record of your care within a health system. An EMR is simply a computerized version of a paper medical record.

If you are receiving care or have received care within the University of Pennsylvania Health System (UPHS) (outpatient or inpatient) and are participating in a University of Pennsylvania research study, results of research-related procedures (i.e., laboratory tests, imaging studies, and clinical procedures) may be placed in your existing EMR maintained by UPHS.

Once placed in your EMR, these results are accessible to appropriate UPHS workforce members that are not part of the research team. Information within your EMR may also be shared with others who are determined by UPHS to be appropriate to have access to your EMR (e.g., health insurance company, disability provider).

## What information about me may be collected, used, or shared with others?

The following personal health information will be collected, used for research, and may be disclosed during your involvement with this research study:

- Personal medical history
- Current and past medications or therapies
- Information from a physical examination that generally also includes your weight, blood pressure reading, heart rate, breathing rate and temperature
- Results of tests and procedures you will undergo during this research study as described in the informed consent form.
- Social security number for the purpose of reimbursement for certain expenses such as parking
- Medical record number
- Any other unique identifying number (such as study ID number linked with your medical records in a separate research file)
- Dates directly related to you, such as your birthdate, dates of hospitalizations, tests, and procedures
- Name, telephone number, fax number, and email addresses may be collected in order to contact you

## Why is my information being used?

Your information is used by the research team to contact you during the study. Your information and results of tests and procedures are used to:

- Do the research
- Oversee the research
- To see if the research was done the right way.

## Who may use and share information about me?

The following individuals may use or share your information for this research study:

- The Principal Investigators and the Investigators' study team
- Authorized members of the workforce of the UPHS and the School of Medicine, and University of Pennsylvania support offices, who may need to access your information in the performance of their duties (for example: for research oversight and monitoring, to provide treatment, to manage accounting or billing matters, etc.).

## Who, outside of the School of Medicine, might receive my information?

As part of the study, the Principal Investigator, the study team and others listed above, may disclose your personal health information, including the results of the research study tests and procedures. This information may be disclosed to those listed below:

### <u>Individuals or organizations responsible for administering the study:</u>

- Your information will be sent to Merck, its authorized representatives, and the FDA.
   Merck and its study representatives monitoring the study will periodically review
   medical and research records to insure integrity of the data being collected. Your
   information will also be sent to labs performing analyses for the study.
- All research centers participating in the study, even if they are not a part of the School of Medicine, may receive information about your medical record but this information will not include any confidential identifying information about you.

## Regulatory and safety oversight organizations

- The Food and Drug Administration
- The Office of Human Research Protections

Once your personal health information is disclosed to others outside the School of Medicine, it may no longer be covered by federal privacy protection regulations.

The Principal Investigators or study staff will inform you if there are any additions to the list above during your active participation in the trial. Any additions will be subject to University of Pennsylvania procedures developed to protect your privacy.

### City of Philadelphia Health Department/PA Department of Health

If you test positive for Hepatitis C, by law we have to report the infection to the City of Philadelphia Health Department/PA Department of Health. We would report your name, gender, racial/ethnic background, and the month and year you were born. This is to keep track of how many people in the U.S. have HCV infection. It is also to make sure that states get enough money from the federal government to support the medical care of people living with HCV. The Health Department does not share the names of HCV infected people with anyone else. It removes all personal identifiers, such as your name, before giving information on the number of HCV infections to the federal government.

# How long may the School of Medicine use or disclose my personal health information?

Your authorization for use of your personal health information for this specific study does not expire.

Your information may be held in a research database. However, the School of Medicine may not re-use or re-disclose information collected in this study for a purpose other than this study unless:

- You have given written authorization
- The University of Pennsylvania's Institutional Review Board grants permission
- As permitted by law

# Can I change my mind about giving permission for use of my information?

Yes. You may withdraw or take away your permission to use and disclose your health information at any time. You do this by sending written notice to the investigators for the study. If you withdraw your permission, you will not be able to stay in this study.

## What if I decide not to give permission to use and give out my health information?

Then you will not be able to be in this research study. You will be given a copy of this Research Subject HIPAA Authorization describing your confidentiality and privacy rights for this study.

By signing this document, you are permitting the School of Medicine to use and disclose personal health information collected about you for research purposes as described above.

# Who can I call with questions, complaints or if I'm concerned about my rights as a research subject?

If you have questions, concerns or complaints regarding your participation in this research study or if you have any questions about your rights as a research subject, you should speak with the Principal Investigators listed on page one of this form. If a member of the research team cannot be reached or you want to talk to someone other than those working on the study, you may contact the Office of Regulatory Affairs with any question, concerns, or complaints at the University of Pennsylvania by calling (215) 898-2614.

When you sign this form, you are agreeing to take part in this research study. This means that you have read the consent form, your questions have been answered, and you have decided to volunteer. Your signature also means that you are permitting the University of Pennsylvania to use your personal health information collected about you for research purposes within our institution. You are also allowing the University of Pennsylvania to disclose that personal health information to outside organizations or people involved with the operations of this study.

| A copy of this consent form will be giv | ren to you. | |
|------------------------------------------|----------------------|------|
| Printed Name of Subject | Signature of Subject | Date |
| Printed Name of Person Obtaining Consent | Signature | Date |

## **Stored Samples and Future Research (Optional)**

If you agree to participate in this study, you may also agree to let us store your samples for future research. These stored samples may help us learn more about hepatitis C. We will label your stored samples with a code that only the study team can link to you. We will keep any information that can be traced back to you as private as possible. If you change your mind and decide you do not want us to store your samples, please contact us. We will do our best to comply with your request, but cannot guarantee that we will always be able to destroy all your samples.

We might send your samples to other investigators for their research, without any information that can identify you. We might also share information such as your sex, age, health history, or ethnicity. We will not sell your samples and you will not be paid for any products that result from the research. Some future studies may need health information (such as smoking history or present health status) that we don't already have. If so, our study team will contact you. Future research that uses your samples will probably not help you, but it may help us learn more about how to treat or prevent hepatitis C and other health problems. In general, the research tests we perform are not like routine medical tests, and may not relate directly to your medical care.

| 1 1 | Check box if you are willing to allow the study team to take and store a sample of your blood for future genetic testing. | |
|---|---|---|
| samples with other rese | ling to allow the study team to sharch teams to learn about hepat<br>I, would not be labelled with you | itis C virus. The |
| Printed Name of Subject | Signature of Subject | Date |
| Printed Name of Person Obtaining Consent | Signature | Date |

## FORMULARIO DE AUTORIZACIÓN EN VIRTUD DE HIPAA (LEY DE TRANSFERENCIA Y RESPONSABILIDAD DE LOS SEGUROS DE SALUD) Y CONSENTIMIENTO INFORMADO PARA SUJETOS DE INVESTIGACIÓN DE LA UNIVERSIDAD DE PENSILVANIA

| Título del protocolo: | Estudio abierto de Zepatier para el tratamiento de pacientes que no padecen de hepatitis C y reciben trasplantes cardíacos de donantes que padecen de hepatitis C (USHER) |
|---|---|
| Patrocinador: | Universidad de Pensilvania (University of Pennsylvania) |
| Proveedor de fondos: | Merck & Co. |
| Investigador principal: | David Goldberg, MD, MSCE (215) 746-8598 |
| Coinvestigador principal: | Peter Reese, MD, MSCE<br>(215) 900-3782<br>Rhondalyn Forde-McLean, MD, MHS<br>(215) 662-2727 |
| Coordinadora del estudio: | Anna Sicilia, BS<br>(215) 746-7105 |
| Contacto de emergencia: | Números de teléfono de emergencia las 24 horas<br>Dr. Reese: (215) 900-3782 Dr. Goldberg: (646) 242-6349<br>(215) 662-6200. Solicite hablar con el coordinador de trasplante<br>cardíaco de guardia. |

## ¿Por qué me solicitan ser voluntario?

Se le solicita que participe en este estudio debido a que se estima que usted debe esperar de 6 a 12 meses o más para recibir un trasplante cardíaco.

Le solicitamos que considere participar en un estudio en el que se ofrecerán corazones con hepatitis C a personas como usted, que no tienen hepatitis C. La hepatitis C es un virus que infecta el hígado, y en el transcurso de muchos años (de 10 a 30) puede causar fibrosis cicatricial hepática y derivar en fibrosis hepática en fase terminal (llamada "cirrosis"), lo que podría ocasionar insuficiencia hepática, cáncer o la muerte. En raras ocasiones, la hepatitis C puede causar inflamación en otras partes del cuerpo, incluso en la piel o en los riñones.

Si usted recibiera un corazón con hepatitis C, le daríamos medicamentos gratis para tratar el virus de la hepatitis C. Los tratamientos para la hepatitis C son sumamente eficaces. En otros estudios, estos medicamentos han curado a más del 95 % de los

pacientes con hepatitis C crónica. Sin embargo, no sabemos si esos medicamentos serán tan eficaces para una persona que se infecta con hepatitis C después de un trasplante cardíaco.

Su participación es voluntaria, lo que significa que usted puede decidir si desea participar o no. Si decide no participar, su atención en Penn y su prioridad en la lista de espera de trasplante cardíaco no se verán afectadas. Recibirá el tratamiento habitual para una persona que se encuentra en la lista de espera de un trasplante.

Antes de tomar su decisión, necesitará saber de qué se trata el estudio, los posibles riesgos y beneficios de participar en este estudio, y qué tendrá que hacer durante el estudio. El equipo de investigación hablará con usted sobre el estudio de investigación y le solicitarán que lea con atención este formulario de consentimiento. También puede decidir conversarlo con su familia, sus amigos y su médico de cabecera. Es posible que algunos términos médicos le resulten difíciles de entender. Pregúntele al médico del estudio o al equipo de investigación sobre el contenido de este formulario. Si decide participar, se le solicitará que firme este formulario.

## ¿Cuál es el propósito de este estudio de investigación?

Actualmente, hay más de 4000 personas en los Estados Unidos que esperan un trasplante cardíaco, pero solo se realizan 2800 trasplantes cardíacos por año con donantes fallecidos. Debido a que no hay suficientes corazones disponibles para todas las personas que los necesitan, el tiempo de espera promedio para un trasplante cardíaco puede ser de 6 a 12 meses o más, especialmente para pacientes con grupos sanguíneos A, B u O, o para pacientes de más estatura o peso.

Una posible opción para aumentar la cantidad de corazones disponibles es permitirles a los pacientes sin hepatitis C aceptar un corazón de un donante con hepatitis C. En la mayoría de los casos, los corazones de donantes con hepatitis C no se dan a pacientes sin hepatitis C.

El propósito de este estudio es determinar si es seguro dar un corazón de un donante con hepatitis C a un receptor sin hepatitis C. Además, este estudio evaluará si los tratamientos administrados después del trasplante pueden curar la hepatitis C en personas que han recibido el corazón de un donante con hepatitis C.

En este estudio, a las personas que reciban un corazón infectado con hepatitis C se les dará como tratamiento un comprimido de grazoprevir + elbasvir (Zepatier) después del trasplante. Esos dos medicamentos combinados en un comprimido han recibido recientemente la aprobación de la Administración de Alimentos y Medicamentos (Food and Drug Administration, FDA) en los EE. UU. para el tratamiento de la hepatitis C crónica en adultos.

Este estudio está financiado por Merck, la compañía que elabora Zepatier.

# ¿Cuánto tiempo tendré que participar en el estudio? ¿Cuántos participantes habrá en el estudio?

Los participantes permanecerán en el estudio durante el tiempo de espera de un trasplante cardíaco (se estima un período aproximado de 3 a 6 meses, pero puede ser más breve o más prolongado) y durante aproximadamente 1 año después de haber

recibido el trasplante, a fin de permitir el seguimiento de su estado de salud antes y después del trasplante. Una vez que los sujetos reciban un trasplante cardíaco de un donante con hepatitis C, se les realizará un seguimiento hasta que su nivel de hepatitis C sea positivo. En ese momento comenzará el tratamiento para la hepatitis C, que durará entre 12 y 16 semanas según el subtipo específico del virus de la hepatitis C que tengan.

En este estudio se inscribirá aproximadamente a 30 pacientes en el Hospital de la Universidad de Pensilvania (Hospital of the University of Pennsylvania, HUP). Prevemos que, de esos 30 pacientes, diez recibirán un trasplante de corazón con hepatitis C. Consideramos que todos los pacientes que reciban un trasplante se infectarán con el virus de la hepatitis C y, por consiguiente, necesitarán tratamiento para el virus de la hepatitis C.

## ¿Qué me piden que haga?

Su participación en el estudio implicará varias visitas al Hospital de la Universidad de Pensilvania durante un período de hasta 6 meses después del trasplante cardíaco (cada visita del estudio generalmente coincidirá con una visita habitual posterior al trasplante cardíaco), y una visita adicional a los 12 meses de haber recibido el trasplante cardíaco. Mientras usted esté en la lista de espera, también controlaremos su estado de salud. Muchas de esas visitas requerirán la obtención de sangre para realizar análisis de seguridad (como análisis de sangre y hepáticos) y análisis para determinar el nivel del virus de la hepatitis C en la sangre (carga viral de la hepatitis C), así como pruebas especiales con ultrasonido para medir la rigidez del hígado.

## Este estudio comprende tres (3) fases:

### Fase 1: Selección

En el período de selección se determina si usted reúne los requisitos necesarios para participar en el estudio. Esta fase tiene lugar antes de que usted reciba un trasplante de corazón con hepatitis C y antes de que comience el tratamiento con el medicamento del estudio. En la selección, usted deberá leer y firmar este consentimiento antes de iniciar cualquier procedimiento del estudio. Es posible que ya le hayan hecho algunos de los exámenes, análisis o procedimientos como parte de su atención habitual. Si ya le han hecho algunos de esos estudios, es posible que no tengan que repetirse. La decisión dependerá del médico del estudio. Los procedimientos de la selección pueden durar hasta 5 horas e incluyen lo siguiente:

- Un examen físico completo.
- Revisión de los medicamentos.
- Evaluación del estado actual de salud.
- Obtención de muestras de sangre:
  - para medir los recuentos sanguíneos y evaluar la función de órganos como el corazón y el hígado;
  - para una prueba de embarazo (en las mujeres que pueden tener hijos);
  - con fines de investigación (esto podría incluir análisis para evaluar las respuestas inmunitarias).

## Fase 2: Lista de espera

Después de la selección, si se determina que usted cumple con los requisitos necesarios para participar en el estudio, modificaremos sus registros de trasplante para establecer que usted acepta y es elegible para recibir ofrecimientos de corazones de donantes con hepatitis C. Usted permanecerá en la lista de espera para el trasplante cardíaco. Durante ese período, aún podrá recibir ofrecimientos de corazones de donantes sin hepatitis C.

Si recibe el ofrecimiento de un corazón con hepatitis C, haremos análisis para determinar el genotipo de la hepatitis C del donante. Solamente aceptamos corazones de donantes que tengan los genotipos 1 y 4 de hepatitis C, porque esos tipos del virus de la hepatitis C son más fáciles de tratar. El análisis del genotipo de la hepatitis C no es totalmente exacto; sin embargo, los estudios han demostrado que tiene una precisión >95 %. No obstante, todos los genotipos de la hepatitis C pueden tratarse, aunque algunos genotipos son más difíciles de tratar que otros (pero con los tratamientos disponibles en la actualidad, pueden lograrse tasas de curación de aproximadamente el 90 % con todos los genotipos).

Si usted recibe el ofrecimiento de un corazón, puede decidir con el médico si desea aceptarlo o no.

Si usted no recibe un trasplante cardíaco de un donante con hepatitis C durante el período del estudio, o si recibe un trasplante de corazón sin hepatitis C, no necesitará ningún tratamiento relacionado con el estudio ni ninguna visita del estudio relacionada con el tratamiento. Revisaremos sus registros médicos para controlar su salud.

Si recibe un trasplante de corazón con hepatitis C, deberá asistir a las visitas del estudio que tienen lugar el mismo día que su visita habitual con el médico. Supervisaremos con atención su estado de salud. Si detectamos el virus de la hepatitis C en su sangre, le daremos un tratamiento para la infección. En ese momento ingresará a la fase 3 del estudio, que se describe a continuación.

#### Fase 3: Trasplante

Le controlaremos la sangre para detectar la infección por hepatitis C. Es posible que algunas personas infectadas con hepatitis C por un trasplante cardíaco puedan eliminar el virus por sí solas mediante el sistema inmunitario. Sin embargo, prevemos que casi todas las personas del estudio que reciban un trasplante de corazón infectado con hepatitis C se infectarán con el virus de manera crónica. Iniciaremos el tratamiento para la hepatitis C tan pronto como detectemos el virus en su sangre.

### Medicamento del estudio

Después del trasplante, los participantes del estudio que tengan hepatitis C recibirán un tratamiento de 12 semanas con Zepatier. El medicamento del estudio consiste en grazoprevir + elbasvir y se administra en un único comprimido combinado por día. En cada visita, le proporcionaremos una cantidad suficiente del medicamento del estudio para que le dure hasta su próxima visita. Asimismo, antes de comenzar con el medicamento, le haremos un control para determinar si hubo mutaciones del virus. Si se hallan ciertas mutaciones, su tratamiento podría extenderse hasta 16 semanas en

lugar de 12, y además recibirá un medicamento adicional, ribavirina, si su función cardíaca lo permite.

Si la hepatitis C no se cura tras haber recibido Zepatier durante 12 semanas, recibirá un segundo tratamiento que incluye Zepatier más 2 medicamentos adicionales que se utilizan para tratar la hepatitis C (sofosbuvir y ribavirina) a fin de curar la infección por hepatitis C.

Zepatier actúa evitando que el virus de la hepatitis C se multiplique en el organismo. En estudios de pacientes con hepatitis C que no han recibido un trasplante cardíaco, las tasas de curación con dichos medicamentos han sido superiores al 95 %.

El medicamento será provisto por el fabricante que patrocina el estudio.

La tasa de curación de Zepatier no se ha establecido en pacientes que se someten a un trasplante cardíaco y se infectan con hepatitis C por el corazón. Tampoco se ha estudiado la seguridad y tolerabilidad de Zepatier después de un trasplante cardíaco. Sin embargo, en caso de que necesite diálisis después del trasplante debido a una insuficiencia renal aguda, sabemos que las tasas de curación en pacientes con hepatitis C y enfermedad renal crónica (incluso en diálisis) conocidas son similares a las tasas de pacientes sin enfermedad renal.

Zepatier ha sido aprobado por la Administración de Alimentos y Medicamentos (FDA). Se eligió este régimen farmacológico como tratamiento de primera línea para este estudio, en lugar de otros medicamentos aprobados, debido a que este medicamento en investigación es único en cuanto a que puede usarse de manera segura en pacientes con funcionamiento cardíaco anormal. En consecuencia, si su funcionamiento cardíaco no se ha recuperado plenamente al inicio del tratamiento después del trasplante, podrá recibir de manera segura los medicamentos en investigación.

#### Otros medicamentos

Durante el estudio, seguirá tomando todos los otros medicamentos indicados por el médico. En la visita de selección, se revisará la lista de medicamentos que toma y se aprobará si usted cumple con los requisitos necesarios para participar en el estudio. Es sumamente importante que en cada visita proporcione la lista exacta de todos los medicamentos que toma (con receta, de venta libre y de hierbas) y que tome su medicación según lo indicado. Sin embargo, <u>no</u> proporcionaremos otros medicamentos.

**Visitas 1 a 4 del estudio:** La primera visita tendrá lugar en el hospital durante su recuperación de la cirugía. Las visitas 2 a 4 tendrán lugar aproximadamente cada semana, los mismos días que sus visitas a la clínica por el trasplante cardíaco.

Un integrante del equipo de investigación intentará comunicarse con usted antes de cada cita para recordarle dónde debe ir y proporcionarle las instrucciones especiales que correspondan.

Durante esas visitas, es probable que se realice lo siguiente:

 Flebotomía (obtención de una muestra de sangre), para medir la presencia del virus de la hepatitis C y determinar si hubo mutaciones del virus (análisis de resistencia a NS5A), lo que podría requerir un tratamiento más prolongado.

- Los análisis de resistencia a NS5A son un tipo de análisis de sangre para detectar mutaciones del virus. Este análisis no está aprobado por la Administración de Alimentos y Medicamentos (FDA), pero está validado por las Enmiendas para la Mejora de los Laboratorios Clínicos (Clinical Laboratory Improvement Amendments, CLIA). Las CLIA son una certificación que permite que los resultados de los laboratorios clínicos se compartan con los pacientes. Este análisis es parte de la atención clínica de rutina, y está recomendado por la FDA para que se utilice con el fin de orientar las decisiones sobre el tratamiento en pacientes con hepatitis C de genotipo 1a (un subtipo del genotipo 1) que reciben tratamiento con Zepatier.
- Le preguntarán cómo se siente y le realizarán un examen físico, si es necesario.
- Revisión de sus medicamentos.

Si los análisis de sangre demuestran que usted tiene hepatitis C, lo llamaremos y haremos arreglos para que inicie el tratamiento contra la hepatitis C. También le notificaremos a su equipo médico que usted va a comenzar el tratamiento contra la hepatitis C.

**Visitas 5 a 9 del estudio:** Estas visitas tendrán lugar aproximadamente cada dos a cuatro semanas, los mismos días que sus visitas a la clínica por el trasplante cardíaco.

Un integrante del equipo de investigación intentará comunicarse con usted antes de cada cita para recordarle a dónde debe ir y proporcionarle las instrucciones especiales que correspondan.

Es posible que, entre las citas, reciba llamadas telefónicas del personal de investigación para confirmar que usted está tomando el medicamento del estudio según lo indicado.

Es probable que se realicen los siguientes procedimientos:

- Obtención de muestras de sangre para medir la presencia del virus de la hepatitis C.
- Le preguntarán cómo se siente y le realizarán un examen físico, si es necesario.
- Revisión de sus medicamentos.
- Evaluación de efectos secundarios y posibles eventos adversos.
- Recuento de los comprimidos del medicamento del estudio y revisión del registro diario de medicamentos, con fines de cumplimiento.
- Provisión de comprimidos adicionales del medicamento del estudio.

**Muestras de sangre con fines de investigación:** Durante todo el estudio, obtendremos muestras de sangre para medir la presencia del virus de la hepatitis C. Esto se coordinará con los análisis de sangre para el equipo de trasplante.

**Visitas adicionales:** Las visitas adicionales solo serán necesarias si el tratamiento no cura la hepatitis C. En ese caso, le proporcionaremos Zepatier durante 12 semanas adicionales, y añadiremos otros dos medicamentos para la hepatitis C (sofosbuvir y ribavirina), provistos por los investigadores del estudio. Esos dos medicamentos adicionales deberían aumentar las probabilidades de curar la hepatitis C.

### Período de seguimiento

El período de seguimiento comenzará cuando usted haya dejado de tomar el medicamento del estudio. Es importante que asista a todas las visitas de seguimiento para que puedan revisar su estado de salud.

**Visita 10 del estudio:** Tendrá lugar 6 meses después del trasplante. Es probable que se realicen los siguientes procedimientos:

- Obtención de muestras de sangre.
- Revisión de sus medicamentos.
- Evaluación de efectos secundarios y eventos adversos.
- Evaluación del estado de salud actual.
- Elastografía de transición (FibroScan®).

Durante esta visita, se analizarán con usted los resultados del estudio y, a medida que los resultados de sus análisis estén disponibles, un integrante del equipo del estudio lo mantendrá al corriente sobre el estado de la infección por hepatitis C después del tratamiento.

**Visita 11 del estudio:** Tendrá lugar aproximadamente 12 meses después del trasplante. Es probable que se realicen los siguientes procedimientos:

- Obtención de muestras de sangre.
- Revisión de sus medicamentos.
- Evaluación del estado de salud actual.
- Elastografía de transición (FibroScan®).

## ¿Cuáles son los posibles riesgos o molestias?

El riesgo principal de este estudio es que usted se infecte con hepatitis C. El posible beneficio principal de este estudio es que usted podría recibir un trasplante cardíaco con menos demora que si solo aceptara ofrecimientos de donantes sin hepatitis C.

## 1. <u>Riesgos relacionados con el trasplante de un corazón con hepatitis C</u> Problemas hepáticos

Usted debe saber que es posible que el tratamiento para la hepatitis C después de un trasplante no sea tan efectivo como lo ha sido en pacientes que no tienen un trasplante. También es posible que, después del trasplante cardíaco, la infección por hepatitis C le cause problemas graves de salud, que incluyen insuficiencia hepática o la muerte. En raras ocasiones, la hepatitis C puede causar inflamación hepática grave durante las primeras semanas o meses posteriores a la infección, u ocasionar fibrosis e insuficiencia hepática después de muchos años.

A corto plazo, la infección por hepatitis C puede causar una enfermedad similar a la gripe, que causa fatiga, náuseas, fiebre, dolor abdominal, vómitos, dolor en las articulaciones e ictericia (piel amarillenta). En muy raras circunstancias, la infección

aguda por hepatitis C puede ocasionar inflamación hepática grave o, incluso, insuficiencia hepática, incluido un trastorno llamado "hepatitis colestásica fibrosante". Se desconoce el riesgo de padecer esta complicación en pacientes sin hepatitis C que reciben un trasplante de un donante con hepatitis C. En algunos casos, esta complicación puede tratarse y curarse con los medicamentos que le proporcionarán los investigadores.

La insuficiencia hepática puede ocasionar hinchazón de las piernas, piel amarillenta, sensación molesta de picazón, sangrado, problemas respiratorios y acumulación de líquido en el abdomen. La insuficiencia hepática también puede causar la muerte. Sobre la base de los datos limitados disponibles, consideramos que sería inusual que un participante del estudio presentara insuficiencia hepática en los primeros meses posteriores al trasplante, mientras esté recibiendo el tratamiento que nosotros proporcionamos. Sin embargo, dada la posibilidad de una insuficiencia hepática, solamente inscribimos en este estudio a personas que podrían ser posibles receptoras de un trasplante de hígado en caso de que presentaran insuficiencia hepática después de un trasplante cardíaco; además, un médico especialista en el hígado (hepatólogo) y un cirujano de trasplantes hepáticos le realizarán una evaluación clínica que no se requiere para un trasplante cardíaco.

Si la hepatitis C no puede curarse con los tratamientos de primera y de segunda línea durante este estudio, al cabo de muchos años podría producirse una inflamación continua y fibrosis cicatricial del hígado, que con el trascurso de muchos años puede derivar en cirrosis y, posteriormente, en insuficiencia hepática. La infección por hepatitis C a largo plazo aumenta el riesgo de cáncer de hígado, de insuficiencia hepática que requiere un trasplante de hígado, o de muerte.

### Riesgos adicionales de la hepatitis C:

La hepatitis C puede causar otros tipos de inflamación en el cuerpo, como artritis, erupción, anemia y daño inflamatorio en el corazón trasplantado. Sin embargo, esos problemas deben responder a un tratamiento eficaz para el virus.

También podría existir un pequeño riesgo de que se presente glomeruloesclerosis focal y segmentaria (Focal and Segmental Glomerulosclerosis, FSGS) después de recibir un riñón de un donante con hepatitis C. La FSGS es una enfermedad que daña los filtros del riñón y provoca la pérdida de proteína en la orina. Sin embargo, esta enfermedad también puede presentarse en pacientes que no tienen hepatitis C. A largo plazo, la FSGS puede causar insuficiencia renal. Después del trasplante, controlamos a todos los pacientes para detectar posibles afecciones como la FSGS. También ofreceremos tratamientos para la FSGS, lo que puede ayudar a algunos pacientes.

## Riesgos del análisis utilizado para determinar el genotipo del virus de la hepatitis C

En este estudio, solamente trasplantamos órganos de pacientes con un determinado tipo de hepatitis C: la de genotipo 1. Ese tipo del virus es más fácil de curar. Existe una probabilidad inferior al 1 % de que el análisis que utilicemos para identificar el virus no tenga una precisión del 100 %. Si el análisis arroja un resultado erróneo y

usted recibe un corazón con un genotipo diferente del virus, las probabilidades de cura podrían ser menores.

## 2. <u>Riesgos relacionados con el medicamento del estudio</u> Efectos secundarios del medicamento:

Cuando reciba tratamiento para la hepatitis C, es posible que sufra efectos secundarios. Se controlará rigurosamente a todos los participantes del estudio para detectar posibles efectos secundarios. Los efectos secundarios pueden ser leves o graves. Debe hablar con el médico del estudio sobre cualquier efecto secundario que usted presente durante su participación en el estudio. Si se lesiona por alguna razón durante su participación en el estudio, debe comunicarle al médico o al hospital tratante que usted está participando en el estudio.

## Efectos secundarios de Zepatier

Si se toman medicamentos que no son del estudio junto con el medicamento del estudio, existe el riesgo de que se presenten efectos secundarios graves o que pongan en riesgo la vida. Por su seguridad, infórmele al médico del estudio o al enfermero del estudio todos los medicamentos que está tomando antes de comenzar a tomar el medicamento del estudio y antes de tomar cualquier otro medicamento durante su participación en el estudio. Asimismo, debe informarle al médico del estudio o al enfermero del estudio antes de inscribirse en otros ensayos clínicos durante su participación en este estudio.

En los estudios, este medicamento ha sido bien tolerado en general. Los riesgos y efectos secundarios relacionados con Zepatier incluyen los siguientes:

#### Muy frecuentes

1) Sensación de cansancio o debilidad, 2) dolor de cabeza.

#### Menos frecuentes

3) Náuseas, 4) diarrea, 5) insomnio, 6) dolor en las articulaciones, 7) prurito 8) erupción, 9) dificultad para respirar, 10) anemia (bajo recuento de glóbulos rojos).

## Muy poco frecuentes

11) Pruebas de la función hepática anormales que sugieren inflamación del hígado, 12) pruebas de la función pancreática anormales que sugieren inflamación del páncreas, 13) depresión, 14) dolor abdominal, 15) irritabilidad.

Infórmele de inmediato a su proveedor de salud si tiene alguno de los siguientes síntomas o si empeoran durante el tratamiento con Zepatier:

- pérdida del apetito;
- color amarillento en la piel o en los ojos;
- náuseas y vómitos;
- cambio de color en las heces;
- sensación de cansancio o debilidad.

Podría haber otros efectos secundarios que aún no se han señalado, incluida una reacción alérgica grave. También es posible que la toma de medicamentos para evitar que el sistema inmunitario rechace el trasplante cardíaco (también denominado "inmunosupresión") junto con Zepatier modifique la eficacia o los efectos secundarios de este medicamento.

## Resistencia del virus a los tratamientos para la hepatitis C:

Desconocemos el grado de eficacia de Zepatier para eliminar el virus de la hepatitis C después de un trasplante, en sus circunstancias. Determinar la eficacia de los medicamentos es uno de los propósitos de nuestro estudio. Uno de los riesgos principales de participar en este estudio es la posibilidad de que la hepatitis C sea resistente a los medicamentos y pueda limitar sus futuras opciones de tratamiento. La probabilidad de que se produzca una resistencia es mayor si se saltea una dosis o si no sigue las recomendaciones del estudio. Si usted demuestra una posible resistencia al medicamento del estudio al presentar un incremento en la carga viral de la hepatitis C, se le solicitará que se vuelva a realizar el análisis de carga viral de la hepatitis C cuanto antes. Podríamos cambiar su plan de tratamiento.

Muy pocas personas (aproximadamente el 5 %) tienen una mutación de un tipo de hepatitis C que presenta riesgo de resistencia. Llevaremos a cabo un análisis para determinar si usted tiene dicho riesgo. Tal como ocurre con el análisis del genotipo, existe un riesgo de que el análisis no tenga una exactitud del 100 %. Si el análisis arroja un resultado erróneo, las probabilidades de cura podrían ser menores y es posible que necesite tratamiento adicional.

Si no responde al tratamiento con Zepatier después de 12 semanas, le ofreceremos un conjunto de medicamentos diferentes (sofosbuvir y ribavirina) además de otro régimen de tratamiento con Zepatier para tratar la hepatitis C. Se desconoce la eficacia de dicho conjunto alternativo de medicamentos para curar la hepatitis C, aunque los investigadores prevén que es probable que cure con eficacia la enfermedad.

Los riesgos y efectos secundarios relacionados con la administración adicional de sofosbuvir y ribavirina incluyen los siguientes:

#### Muy frecuentes

1) Sensación de cansancio o debilidad, 2) dolor de cabeza, 3) náuseas/dolor de estómago, 4) anemia, 5) insomnio, 6) erupción, 7) prurito, 8) dificultad para respirar.

#### Menos frecuentes

9) Tos, 10) piel reseca, 11) diarrea, 12) vómitos, 13) disminución del apetito, 14) indigestión, 15) dolor muscular, 16) irritabilidad/depresión, 17) dolor en las articulaciones, 18) irritación nasal, 19) pruebas de la función hepática anormales, 20) pruebas de la función pancreática anormales, 21) recuento bajo de glóbulos blancos, lo cual podría aumentar la vulnerabilidad a las infecciones, 22) bajo recuento plaquetario, lo cual podría aumentar la vulnerabilidad al sangrado, 23) anomalías congénitas debido a la ribavirina cuando el hombre o la mujer están tomando ribavirina en el momento de la concepción o han tomado ribavirina durante los 6 meses anteriores.

## 3. <u>Riesgos relacionados con los procedimientos y análisis del estudio</u> Extracción de sangre

Los posibles riesgos de la introducción de la aguja para extraer sangre incluyen dolor, hematomas, sangrado, desmayo e infección. Las molestias ocasionadas por este

procedimiento generalmente son breves, y los efectos secundarios graves son extremadamente inusuales. Algunas personas tienen sensación de mareo o vahído tras la extracción de sangre. La cantidad de sangre que se extraiga estará dentro de los límites permitidos para los participantes adultos.

### Pruebas genéticas

Parte de la sangre que le extraigan como parte de este estudio se utilizará para pruebas genéticas. Las pruebas genéticas pueden ayudar a los investigadores a conocer las posibles relaciones entre la respuesta al tratamiento contra el virus de la hepatitis C y los factores genéticos. También se realizará un análisis de antígenos leucocitarios humanos (Human leukocyte antigen, HLA). Es una prueba genética de marcadores del sistema inmunitario.

No divulgaremos ningún tipo de información sobre usted o su familia a parientes, compañías de seguros, empleadores o médicos de atención primaria sin su autorización por escrito. Podría existir el riesgo de que la información genética obtenida como resultado de la participación en la investigación se utilice indebidamente con fines discriminatorios. Sin embargo, las leyes federales y estatales proporcionan algunas protecciones contra la discriminación genética. Los investigadores que tengan acceso a su información genética tomarán medidas para mantener la confidencialidad de dicha información. Si bien tenemos el compromiso de mantener la confidencialidad, un tribunal podría presentar una orden judicial para obtener sus registros médicos. Todas estas cuestiones deben considerarse con mucho cuidado antes de tomar la decisión de participar en el estudio.

## Riesgo de las muestras almacenadas (opcional)

Si usted acepta que se almacenen muestras para investigaciones en el futuro, podría haber riesgos de pérdida de confidencialidad relacionados con el almacenamiento y análisis de sus muestras o de la información obtenida del análisis de sus muestras. Por ejemplo, si una investigación futura incluye pruebas genéticas, existe un posible riesgo relacionado con la divulgación de información privada de salud a pesar de que tomemos todos los recaudos posibles para mantener su confidencialidad.

## Hallazgo de problemas de salud durante la selección

Durante la selección para este estudio, le haremos exámenes y llevaremos a cabo estudios como parte del proceso de selección. Es posible que, al realizar dichos estudios, detectemos problemas de salud que usted desconocía. Si hallamos problemas de salud nuevos, responderemos sus preguntas e intentaremos acordar el tratamiento apropiado en caso de ser necesario. Si se hallan problemas de salud nuevos, es posible que usted no pueda participar en este estudio. También es posible que, según los resultados, usted ya no cumpla con los requisitos necesarios para recibir un trasplante cardíaco.

### Riesgos para la reproducción

Si usted queda embarazada, es posible que Zepatier provoque problemas en el feto. Actualmente se desconocen los riesgos para el feto o el lactante, de modo que las mujeres que están embarazadas o amamantando NO pueden participar en el estudio.

Antes de recibir el medicamento del estudio, todas las <u>mujeres</u> que puedan tener hijos deben realizarse una prueba que demuestre que no están embarazadas, y se les

aconsejará sobre la importancia de evitar el embarazo, que incluye la importancia del uso de métodos anticonceptivos de alta eficacia, durante el tratamiento del estudio. Las mujeres que pueden tener hijos deben adoptar un método anticonceptivo de alta eficacia durante su participación en el estudio y las seis semanas posteriores. Definimos "método anticonceptivo de alta eficacia" del mismo modo en que lo define el programa de trasplante. En particular, la toma de medicamentos para evitar el rechazo del trasplante puede causar anomalías congénitas.

Los ejemplos incluyen los siguientes:

- 1) abstinencia sexual;
- 2) pareja con vasectomía;
- 3) dispositivo intrauterino (DIU);
- 4) un método hormonal, como píldoras anticonceptivas MÁS un método de barrera, como preservativos;
- 5) diafragma con espermicida MÁS preservativo.

Aun si utiliza un método anticonceptivo, existe una pequeña probabilidad de que quede embarazada. Si sospecha que está embarazada, debe informárselo de inmediato al médico del estudio. Si queda embarazada durante su participación en el estudio, es importante que nos informe de inmediato.

<u>Todos los hombres y las mujeres</u> del estudio que sean sexualmente activos deben utilizar TAMBIÉN un método anticonceptivo de barrera, como preservativos, durante su participación en el estudio y mientras tengan hepatitis C. Si bien es inusual, la hepatitis C puede, a veces, contagiarse a través de relaciones sexuales. Es importante usar un anticonceptivo de barrera durante *cualquier* actividad sexual para evitar que su pareja se infecte con el virus.

Todos los hombres y las mujeres que necesiten tratamiento con ribavirina deberán usar dos tipos de métodos anticonceptivos mientras estén en tratamiento y hasta 6 meses después de la última dosis del medicamento del estudio, debido al riesgo de anomalías congénitas por el uso de ribavirina. También se requiere que los hombres usen un método anticonceptivo porque la ribavirina puede afectar los espermatozoides y ocasionar anomalías congénitas.

## ¿Qué ocurrirá si surge información nueva sobre el estudio?

Además de los riesgos antedichos, es posible que existan riesgos que se desconocen, o riesgos no previstos, relacionados con la participación en el estudio. Si surge nueva información sobre el medicamento del estudio que pudiera afectar su decisión de continuar participando, el médico del estudio se lo informará de inmediato y analizará con usted su decisión de continuar participando en el estudio clínico.

Es posible que le soliciten firmar un formulario de consentimiento revisado en caso de que esto ocurra. Usted tiene el derecho de decidir si va a continuar en el estudio clínico o si desea retirarse.

## ¿Cuáles son los posibles beneficios del estudio?

El beneficio principal del estudio es que usted puede recibir un trasplante con menos demora que si decidiera esperar un corazón sin hepatitis C. Recibir un trasplante cardíaco sin esperar tanto brindará beneficios clínicos conforme mejore su

funcionamiento cardíaco y su calidad de vida. Además, recibir un trasplante cardíaco podría aumentar su esperanza de vida al disminuir el riesgo de muerte durante el período de espera del trasplante.

## ¿De qué otras opciones dispongo si no participo?

Recomendamos que converse con su médico sobre este estudio y que analice otras opciones de tratamiento. Las otras opciones de tratamiento incluyen no inscribirse en este estudio y esperar un trasplante de corazón de un donante que no tenga hepatitis C.

Sin embargo, si decide no participar en el estudio, podría seguir en la lista de espera durante un período más prolongado y sufrir consecuencias que afecten su salud, incluidas la muerte o complicaciones adicionales.

## ¿Me pagarán por participar en este estudio?

Usted no recibirá ninguna remuneración por su participación en este estudio.

## ¿Tengo que pagar algo?

El trasplante cardíaco lo pagará su compañía de seguros, y no requiere ninguna autorización previa adicional para la posibilidad de recibir un corazón de un donante con hepatitis C. El costo de todas las visitas, los análisis y los procedimientos antedichos se les cobrará a usted o a su compañía de seguros, excepto la extracción de sangre con fines de investigación (que incluye el análisis del genotipo de la hepatitis C, que se basa en un análisis desarrollado en laboratorio con materiales adquiridos en la entidad comercial que desarrolló el análisis, y que pagará el equipo de investigación) y el medicamento del estudio, que pagará el financiador del estudio. Usted sigue siendo responsable de todos los deducibles o copagos correspondientes a las visitas de rutina en el consultorio, los análisis de sangre y los procedimientos. Hable con el médico y el equipo del estudio para que lo comuniquen con un asesor financiero a fin de determinar exactamente de cuánto será su deducible y su copago; estos montos varían considerablemente según el tipo de seguro.

## ¿Qué sucede si me lesiono por participar en el estudio?

Si usted se enferma o se lesiona como resultado directo de ingerir los productos del estudio, el Hospital de la Universidad de Pensilvania le proporcionará tratamiento médico. El patrocinador, la Universidad de Pensilvania, le reembolsará todos los costos necesarios razonables de dicho tratamiento médico. El patrocinador no ofrece ninguna otra forma de reembolso por enfermedades o lesiones relacionadas con el estudio. En caso de que usted presente una enfermedad o lesión relacionada con el estudio, debe comunicarse de inmediato con el médico del estudio según la información de contacto que figura en la primera página de este formulario.

Si recibe beneficios de Medicare, la ley requiere que el patrocinador, la Universidad de Pensilvania, notifique los pagos que le efectúen a usted por el tratamiento, las complicaciones y las lesiones que pudieran surgir de este estudio. A tales efectos, se les proporcionará a los Centros de Servicios de Medicare y Medicaid, sus agentes o proveedores, la información sobre su participación en el estudio, los tratamientos médicos que recibió, los reclamos de Medicare y otra información personal como su nombre, su número de seguro social y su fecha de nacimiento.

Al firmar este formulario, usted no renuncia a ninguno de sus derechos legales.

Si considera que se ha lesionado como resultado de su participación en este estudio de investigación, infórmeselo cuanto antes a la persona a cargo del estudio de investigación. El nombre y el número de teléfono del investigador figuran al comienzo del formulario de consentimiento.

Tenemos el compromiso de ofrecerle tratamiento para la infección por hepatitis C durante el estudio. Esperamos que dichos tratamientos tengan la probabilidad de curar su infección. Sin embargo, es posible que el tratamiento no cure la infección y que usted presente complicaciones de salud. Una vez que finalice el estudio, esperamos que usted procure tratamientos adecuados para la infección por hepatitis C a través de su seguro médico o en forma privada.

# ¿Cuándo finaliza el estudio? ¿Puedo retirarme del estudio antes de que termine?

Se prevé que este estudio finalice una vez que todos los participantes hayan completado todas las visitas, y que se haya recopilado toda la información. Si está considerando o ha decidido retirarse del estudio, infórmeselo al médico del estudio. Él le dirá cómo retirarse del estudio de manera segura. Si está pensando en retirarse del estudio, es importante que se lo informe al médico del estudio, ya que él podrá evaluar todos los riesgos y analizar qué tipo de atención y análisis de seguimiento alternativos podrían ser los mejores para usted.

### Motivos para interrumpir el medicamento del estudio

Si usted no está respondiendo bien al medicamento del estudio (con controles frecuentes de los niveles de hepatitis C en la sangre) o si presenta una complicación que podría poner en riesgo su vida debido al medicamento, interrumpiremos de inmediato los medicamentos del estudio. No obstante, deberá recibir seguimiento, aunque con menos frecuencia. Independientemente del estado de la enfermedad hepática, la recomendación es tratar la hepatitis C si es posible en términos médicos; sin embargo, algunos médicos podrían elegir esperar y no tratar la enfermedad en el futuro inmediato.

### Motivos para el retiro o la interrupción del estudio

La participación en el estudio depende enteramente de usted. Puede retirarse del estudio en cualquier momento y por cualquier motivo. Si se retira del estudio, su atención futura no se verá afectada. Si decide retirarse del estudio, es posible que le solicitemos que asista a una visita final para realizar análisis y exámenes con motivos de seguridad. Sin embargo, no se le exigirá que asista a dicha visita.

Es posible que lo retiren del estudio sin solicitarle permiso si ocurre lo que se indica a continuación:

 Queda embarazada mientras está siguiendo el tratamiento con Zepatier. Se interrumpirá el tratamiento dado que no existen datos sobre la seguridad de Zepatier durante el embarazo. Las pacientes continuarán con las visitas programadas del estudio, pero no serán elegibles para continuar el tratamiento con Zepatier.

- No podemos localizarlo, falta a varias visitas o se saltea varias dosis del medicamento del estudio.
- Usted presenta un trastorno que pone en peligro su vida o existe otro riesgo significativo según el criterio de los investigadores.
- Según nuestra opinión o la de su proveedor de atención primaria, es mejor para usted que deje de tomar los medicamentos del estudio, aunque no se cumplan los criterios para interrumpir el tratamiento.
- El fabricante deja de elaborar Zepatier, o si se tomó la decisión de dar por terminado el estudio.

# ¿Quiénes pueden ver o utilizar mi información? ¿Cómo se protegerá mi información personal?

Se mantendrá la confidencialidad de sus registros médicos en la medida de lo permitido por la ley. En los informes y publicaciones que se obtengan como resultado de este estudio, no se utilizará su nombre ni ningún otro dato que pudiera identificarlo. Debido a su consentimiento para participar, el patrocinador del estudio o el Comité de Revisión Institucional de la Universidad de Pensilvania ([Penn's Institutional Review Board], el grupo responsable de asegurar que el estudio siga las normas de protección de sujetos humanos de investigación) pueden revisar sus registros médicos con el conocimiento de que dichos registros solamente se utilizarán para el cumplimiento de obligaciones relacionadas con este estudio clínico. También les proporcionaremos información sobre usted a sus médicos personales. Usted puede cambiar de médico cuando lo desee, pero necesitamos tener los datos de un médico con el cual podamos comunicarnos con respecto a usted. No le solicitaríamos su permiso para cada uno de esos contactos.

Los datos de este estudio podrán ingresarse a una base de datos computarizada a través de un sitio web seguro. Solamente se le permitirá el ingreso y el acceso a los datos al personal autorizado, con el uso de una contraseña. En la base de datos del estudio, usted no estará identificado por su nombre, su número de seguro social ni su número de expediente médico. A cada paciente se le asignará un código de identificación único del estudio. El equipo del estudio mantendrá bajo llave los registros que vinculen el código de identificación del estudio con la información de identificación personal.

Según lo exige la ley de los EE. UU., en el sitio web <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a> se encuentra disponible una descripción de este estudio clínico. Dicho sitio web no incluye información que pueda identificarlo a usted. A lo sumo, el sitio web incluirá un resumen de los resultados. Puede realizar búsquedas en ese sitio web en cualquier momento.

## Expedientes médicos electrónicos y resultados de la investigación ¿Qué es un expediente médico electrónico?

Un expediente médico electrónico (Electronic Medical Record, EMR) es una versión electrónica del registro de su atención en un sistema de salud. Un EMR es simplemente una versión computarizada de un expediente médico impreso en papel.

Si usted está recibiendo o ha recibido atención en el Sistema de Salud de la Universidad de Pensilvania (University of Pennsylvania Health System, UPHS), ya sea

como paciente internado o ambulatorio, y se encuentra participando en un estudio de investigación de la Universidad de Pensilvania, los resultados de los procedimientos relacionados con la investigación (es decir, análisis de laboratorio, estudios de imágenes y procedimientos clínicos) podrían incluirse en su EMR existente que mantiene el UPHS.

Una vez ingresados a su EMR, dichos resultados estarán accesibles para los integrantes del personal autorizado del UPHS que no formen parte del equipo de investigación. La información que contiene su EMR también podría compartirse con terceros cuyo acceso a su EMR el UPHS considere apropiado (p. ej., compañías de seguro de salud, proveedores de servicios para discapacitados, etc.).

# ¿Qué información sobre mi persona podría recopilarse, utilizarse y compartirse con terceros?

La siguiente información personal de salud podrá recopilarse, utilizarse para investigación y divulgarse durante su vinculación con este estudio de investigación:

- Historia clínica personal.
- Medicamentos o tratamientos presentes y pasados.
- Información de exámenes físicos, que generalmente incluye su peso, presión sanguínea, frecuencia cardíaca, frecuencia respiratoria y temperatura.
- Resultados de análisis y procedimientos que usted se realizó durante este estudio de investigación, según se describe en el formulario de consentimiento informado.
- Número de seguro social para el reembolso de determinados gastos, como estacionamiento.
- Número de expediente médico.
- Otros números de identificación únicos (como el número de identificación del estudio vinculado a sus registros médicos en un archivo de investigación por separado).
- Datos directamente relacionados con usted, como su fecha de nacimiento, fechas de hospitalizaciones, análisis y procedimientos.
- Podría recopilarse su nombre, número de teléfono, número de fax y dirección de correo electrónico a fin de comunicarse con usted.

## ¿Por qué se utiliza mi información?

El equipo de investigación utiliza su información para comunicarse con usted durante el estudio. Su información y los resultados de los análisis y procedimientos se utilizan para lo siguiente:

- realizar la investigación;
- supervisar la investigación;
- controlar si la investigación se llevó a cabo correctamente.

## ¿Quiénes podrían utilizar y compartir la información sobre mí?

Las siguientes personas podrían utilizar o compartir su información para este estudio de investigación:

• Los investigadores principales y el equipo de estudio de los investigadores.

Integrantes autorizados del personal del UPHS y de la Facultad de Medicina, así
como de las oficinas de apoyo de la Universidad de Pensilvania, quienes podrían
necesitar el acceso a su información para llevar a cabo sus tareas (por ejemplo,
para la supervisión y el control de la investigación, para administrar tratamiento,
para gestionar asuntos contables o de facturación, etc.).

## Fuera de la Facultad de Medicina, ¿quiénes podrían recibir mi información?

Como parte del estudio, el investigador principal, el equipo del estudio y otras personas antedichas podrían divulgar su información personal de salud, incluidos los resultados de los análisis y procedimientos del estudio de investigación. Esta información podría divulgarse a quienes se indican a continuación:

## Personas o entidades responsables de administrar el estudio:

- Su información se enviará a Merck, sus representantes autorizados y la FDA. Merck y sus representantes que supervisan el estudio llevarán a cabo una revisión periódica de los registros médicos y de investigación para garantizar la integridad de los datos que se recopilen. Su información también se enviará a los laboratorios que realicen análisis para el estudio.
- Todos los centros de investigación que participen en el estudio, aunque no formen parte de la Facultad de Medicina, podrían recibir información sobre sus registros médicos, pero dicha información no incluirá ningún dato confidencial de identificación sobre usted.

### Organizaciones de supervisión de la seguridad y de las normas:

- La Administración de Alimentos y Medicamentos (Food and Drug Administration).
- La Oficina de Protección de los Seres Humanos en Investigación (Office of Human Research Protections).

Una vez que su información personal de salud se divulgue a terceros fuera de la Facultad de Medicina, podría dejar de estar cubierta por las normas federales de protección de la privacidad.

Los investigadores principales o el personal del estudio le informarán si se realizan incorporaciones a la lista antedicha durante su participación activa en el ensayo. Todas las incorporaciones estarán sujetas a los procedimientos de la Universidad de Pensilvania desarrollados para proteger su privacidad.

Departamento de Salud de la Ciudad de Filadelfia/Departamento de Salud de Pensilvania (City of Philadelphia Health Department/PA Department of Health):

Si usted obtiene un resultado positivo en el análisis de detección de la hepatitis C, la ley exige que lo notifiquemos al Departamento de Salud de la Ciudad de Filadelfia/Departamento de Salud de Pensilvania (City of Philadelphia Health Department/PA Department of Health). Notificaríamos su nombre, sexo, origen étnico/racial, y el mes y el año de su nacimiento. Esto se realiza para llevar un registro de la cantidad de personas que están infectadas por el virus de la hepatitis C en los EE. UU. También se realiza para garantizar que los estados obtengan dinero suficiente del gobierno federal para mantener la atención médica de las personas con hepatitis C. El Departamento de Salud no comparte con nadie los nombres de las personas

infectadas por el virus de la hepatitis C. Antes de proporcionarle información al gobierno federal sobre la cantidad de infecciones por el virus de la hepatitis C, el Departamento elimina todos los datos de identificación personal, como los nombres.

# ¿Durante cuánto tiempo la Facultad de Medicina puede utilizar o divulgar mi información personal de salud?

Su autorización del uso de su información personal de salud para este estudio específico no tiene vencimiento.

Su información podría mantenerse en una base de datos de investigación. Sin embargo, la Facultad de Medicina podría no volver a utilizar o a divulgar la información recopilada en este estudio con fines que sean distintos a los del estudio a menos que:

- usted otorgue su autorización por escrito;
- el Comité de Revisión Institucional de la Universidad de Pensilvania (University of Pennsylvania's Institutional Review Board) así lo autorice;
- esté permitido por la ley.

# ¿Puedo cambiar de opinión con respecto a mi permiso para que se utilice mi información?

Sí. Usted puede retirar su permiso para usar y divulgar su información de salud en cualquier momento. Debe hacerlo enviando una notificación por escrito a los investigadores del estudio. Si retira su permiso, ya no podrá seguir participando en este estudio.

# ¿Qué sucede si decido no dar mi permiso para usar y divulgar mi información de salud?

En ese caso, ya no podrá seguir participando en este estudio de investigación. Usted recibirá una copia de esta Autorización de la Ley de Transferencia y Responsabilidad de los Seguros de Salud (Health Insurance Portability and Accountability Act, HIPAA) para Sujetos de Investigación que describe sus derechos de privacidad y confidencialidad para este estudio.

Al firmar este documento, usted le permite a la Facultad de Medicina utilizar y divulgar la información personal de salud que se recopiló sobre usted con fines de investigación según lo descrito anteriormente.

## ¿A quién puedo llamar para hacer preguntas o presentar quejas, o si tengo inquietudes sobre mis derechos como sujeto de investigación?

Si tiene preguntas, inquietudes o quejas con respecto a su participación en este estudio de investigación, o si tiene preguntas sobre sus derechos como sujeto de investigación, debe hablar con los investigadores principales, que figuran en primera página de este formulario. Si no puede comunicarse con un integrante del equipo de investigación, o si desea hablar con una persona que no esté trabajando en el estudio, puede hacer preguntas o presentar inquietudes o quejas llamando a la Oficina de Asuntos de Regulación (Office of Regulatory Affairs) de la Universidad de Pensilvania al (215) 898-2614.

Versión 1.5 del Consentimiento/10 de enero de 2018

Al firmar este formulario, usted acepta participar en este estudio de investigación. Esto significa que ha leído el formulario de consentimiento, que se han respondido sus preguntas y que ha decidido participar en forma voluntaria. Su firma también significa que le permite a la Universidad de Pensilvania utilizar la información personal de salud que se recopiló sobre usted con fines de investigación dentro de nuestra institución. Asimismo, le permite a la Universidad de Pensilvania divulgar dicha información personal de salud a organizaciones o personas externas involucradas en las operaciones de este estudio.

| Se le proporcionará a usted una copia | a de este consentimiento informad | 0. |
|---|---|---|
| Nombre del sujeto en letra de imprenta | Firma del sujeto | Fecha |
| Nombre de la persona que obtiene | Firma | Fecha |

## Muestras almacenadas e investigaciones futuras (opcional)

Si usted acepta participar en este estudio, es posible que también acepte permitirnos almacenar sus muestras para investigaciones futuras. Esas muestras almacenadas podrían ayudarnos a conocer más sobre la hepatitis C. Rotularemos sus muestras almacenadas con un código que solamente el equipo del estudio podrá vincular con usted. Mantendremos la privacidad de toda información que pueda identificarlo a usted tanto como sea posible. Si cambia de opinión y decide que dejemos de almacenar sus muestras, comuníquese con nosotros. Haremos todo lo posible por cumplir con su solicitud, pero no siempre podemos garantizar la destrucción total de todas sus muestras.

Podemos enviarles sus muestras a otros investigadores con fines de investigación, sin ninguna información que pueda identificarlo. También podemos compartir información como su sexo, edad, historia clínica u origen étnico. No venderemos sus muestras y no recibiremos pago alguno por los productos que se obtengan como resultado de la investigación. Algunos estudios futuros podrían requerir información de salud (como antecedentes de tabaquismo o estado de salud actual) que actualmente no poseemos. En ese caso, el equipo del estudio se comunicará con usted. Las investigaciones futuras que utilicen sus muestras probablemente no sean útiles para usted, pero podrían ayudarnos a obtener más conocimientos sobre cómo tratar o prevenir la hepatitis C y otros problemas de salud. En general, los análisis de investigación que llevamos a cabo no son como los análisis médicos de rutina, y podrían no estar directamente relacionados con su atención médica.

| · · · · | Marque la casilla si desea permitir que el equipo del estudio obtenga y almacene una muestra de sangre suya para futuras pruebas genéticas. | |
|---|---|---|
| muestras de sangre con conocimientos sobre el conocimiento sobre el conocimientos sobre el conocimiento sobre el | ea permitir que el equipo d<br>n otros equipos de investiga<br>virus de la hepatitis C. Las<br>ularán con su información | ación para obtener más<br>muestras de sangre, si |
| Nombre del sujeto en letra de imprenta | Firma del sujeto | Fecha |
| Nombre de la persona que obtiene el consentimiento en letra de imprenta | Firma | Fecha |